CLINICAL TRIAL: NCT05394948
Title: Design of Healthy and Sustainable Food and Ingredients Based on the Application of the Circular Economy
Brief Title: Circular Economy and the Design of Healthy and Sustainable Food and Ingredients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALISSEC
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2023-01

CONDITIONS: Overweight; Sustainability; Food; Microbiota; Habits
Keywords: Overweight; Microbiota; Sustainability; New food; Food ingredients
MeSH Terms: conditions — Overweight; Habits

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving dietary recommendations including experimental nutraceutic. (Experimental): Experimental group will consume experimental nutraceutic instead of the habitual breakfast during 3 weeks and within a dietary recommendations.
  Interventions: Dietary Supplement: Dietary recommendations including experimental nutraceutic.
- Group receiving dietary recommendations including control nutraceutic. (Active Comparator): Experimental group will consume control nutraceutic instead of the habitual breakfast during 3 weeks and within a dietary recommendations.
  Interventions: Dietary Supplement: Dietary recommendations including control nutraceutic.

INTERVENTIONS:
Dietary Supplement: Dietary recommendations including experimental nutraceutic. — Volunteers allocated in the control group will receive every day and during 3 consecutive weeks the experimental nutraceutic instead of the breakfast. Nutraceutical intake will be accompanied by nutritional advice to follow for the 3 weeks of intervention.
  Arms: Group receiving dietary recommendations including experimental nutraceutic.
Dietary Supplement: Dietary recommendations including control nutraceutic. — Volunteers allocated in the control group will receive every day and during 3 consecutive weeks the control nutraceutic instead of the breakfast. Nutraceutical intake will be accompanied by nutritional advice to follow for the 3 weeks of intervention.
  Arms: Group receiving dietary recommendations including control nutraceutic.

SUMMARY:
There is a need to change eating patterns towards healthier diets with new sources of non-animal protein, obtained through more sustainable systems in line with strategies such as the European Green Deal, the "Farm to Fork" strategy, or the Common Agricultural Policy, among others.

The objective of this study, is to evaluate the nutritional effect of the developed products and their impact on the improvement and/or prevention of health problems (diabetes, intestinal dysbiosis), as well as to design and evaluation of the effect on health of a vegetable protein-based nutraceutical that also includes fiber and resistant starch.

DETAILED DESCRIPTION:
This study is designed as a 3-week, randomised, parallel study, focused on overweight/obese men and women between 20 and 65 years old.

All participants attend the Nutrition Intervention Unit of the Center for Nutrition Research in the University of Navarra for 2 times during the intervention (day 1 and day 21).

RECRUITMENT AND SCREENING:

The recruitment and screening of participants will be carried out through a Google Form questionnaire and by a phone call. At the same time, the database of people interested in participating in nutritional studies of the Center for Nutrition Research will be used, who will be contacted by phone or email to offer them the study. In addition, the study information and the recruitment form will also be posted on the Center for Nutrition Research website for anyone who wants to enroll in the study. On the other hand, the study will be disseminated through the channels available in the University of Navarra (Unclic, Alumni, emails, etc.) and through the placement of informative posters in the different buildings of the University of Navarra, as well as in public and private centers in Navarra, with prior authorization. If it is necessary, the study will be disseminated in the media such as in press, radio and TV.

The staff of the Nutritional Intervention Unit will assess the data provided by the potential participants and those who meet the inclusion criteria will be cited for the first visit of the study, which will take place in the Nutritional Intervention Unit of the Center for Nutrition Research in the University of Navarra. The information sheet and the informed consent will be sent to them beforehand so that they can read it for visit 1.

CLINICAL INVESTIGATION DAY 1 (day 1):

It will be carried out in groups of 10 people, who will attend the facilities of the University of Navarra fasting for at least 10 hours. The volunteers will be received by the nutritionist and the study nurse. Once gathered, proceed as follows:

* Welcome, detailed explanation of the study procedures and resolution of doubts.
* Delivery of the information sheet and the informed consents to the volunteers.
* Those volunteers who want to participate will sign the informed consent. Then, the procedures for taking samples and data will begin.

  * Delivery of 2 kits for collecting stool samples (beginning and end). The sample collected at the beginning will be delivered within three days to the facilities of the Nutritional Intervention Unit.
  * Delivery of a food consumption frequency questionnaire and a gastrointestinal symptoms questionnaire. They will be filled out with the help of the nutritionist during the visit and will refer to the last 3 weeks.
  * Delivery of the VAS hunger-satiety questionnaire to be completed 1-2 days before the final visit.
  * The dietician-nutritionist will take the anthropometric measurements of the volunteers individually and with light clothing.
  * The nurse will draw blood (2 serum tubes of 5 mL).
  * Delivery of the nutraceutical under study or the control nutraceutical (see composition in Table 1) as well as indications for the three weeks of the study. The nutraceutical should be consumed daily for 3 weeks as a substitute for breakfast in both groups.
  * The date and time for the final visit (visit 2) will be specified.

CLINICAL INVESTIGATION DAY 2 (day 21):

It will be carried out in groups of 10 people, who will have to attend the University of Navarra fasting for at least 10 hours. The volunteers will be received by the nutritionist and the study nurse. Once gathered, proceed as follows:

* Collection of stool samples and VAS hunger-satiety questionnaire.
* General talk to welcome everyone and ask about the course of the 3 weeks.
* The dietitian-nutritionist will take the anthropometric measurements of the volunteers individually and with light clothing.
* The Food Frequency Questionnaire and the Gastrointestinal Symptoms Questionnaire corresponding to the final visit will be completed with the help of the nutritionist. They will refer to the 3 weeks that the intervention lasts.
* The volunteer will complete the Nutraceutical Acceptance Questionnaire.
* The nurse will draw blood (2 serum tubes of 5 mL).

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-65 years.
* Body mass index: 25-29.9 kg/m2
* Physical examination and vital signs normal or clinically irrelevant to the experiment.
* Volunteers undergoing pharmacological treatment will be maintained if the dose is stable for at least 3 months before the start of the study, excluding treatments that alter gastrointestinal function, antidiabetics and stomach protectors.
* Subjects must be able to understand and be willing to sign the informed consent, and must comply with all the procedures and requirements of the study.
* Subjects have to present a stable weight (+/-3kg) in the three months prior to the start of the study.

Exclusion Criteria:

* Subjects with relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux, etc.
* Subjects with frecuent flatulence, diarrhea and intestinal discomfort.
* Subjects who have undergone surgical interventions with permanent sequelae in the digestive system (for example, gastroduodenostomy).
* Subjects with a high alcohol intake, more than 14 units (women) and 20 units (men).
* Women who are breastfeeding or pregnant.
* Subjects with liver disease.
* Subjects with some type of cancer or undergoing treatment for it, or who have not had a period of at least 5 years since its eradication.
* Subjects with allergies to any component of the product under study or any other food that interferes and makes it difficult to monitor the study.
* Subjects who present some type of cognitive and/or psychic impairment.
* Subjects in whom poor collaboration is expected or who, in the opinion of the investigator, have difficulties in following the study procedures.
* Subjects who follow some type of supplementation that interferes with the study: probiotics, supplements rich in fiber, laxatives, protein supplements, etc.
* Subjects who are immersed in some treatment for weight loss.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Balanced in men and women.
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change of fecal microbiota from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Fecal microbiota of participants will be analyzed by bacterial 16S gene sequencing technology.

SECONDARY OUTCOMES:
Change of weight from baseline to week 3 (weighing machine) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of body mass index from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Body mass index will be calculated as follows: weight (kg)/ height (cm)2.
Height at baseline. | The Time Frame contains one time point: Clinical Investigation Day 1 (at baseline).
  Height of participants will be measured by stadiometer and reported in meters.
Change of waist circumference from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of glucose concentration from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Change of glucose levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of insulin concentration from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Change of insulin levels of participants in fasting condition will be analyzed by ELISA kit and reported in mU/L.
Change of HOMA index from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Change of HOMA index of participants in fasting condition will be calculated by the following formula: insulin (μU/ml) x glucose (mmol/l)/22,5.
Change of dietary intake from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Change of dietary intake of participants will be analyzed by Food Frequency Questionnaire.
Change of hunger from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  The change in hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of fullness from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  The change in fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of satisfaction from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  The change in satisfaction of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of want to eat something else sensation from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  The change in want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of thirst from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  The change in thirst of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of gastrointestinal symptoms from baseline to week 3. | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 3 weeks of intervention).
  Gastrointestinal symptoms will be analyzed by a gastrointestinal symptom questionnaire.
Nutraceutical acceptance at week 3. | The Time Frame contains Clinical Investigation Day 2 (after 3 weeks of intervention).
  Nutraceutical acceptance will be analyzed by acceptance questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín I Milagro Yoldi, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra. Center for Nutrition Research., Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No